CLINICAL TRIAL: NCT05105646
Title: Are Preoperative Perception of Pain and Psychological Distress Before Primary Knee Arthroplasty Associated With Reason for Revision Surgery? Results of an Observational Study From the Dutch Arthroplasty Register.
Brief Title: Are Perception of Pain and Psychological Distress Before Knee Arthroplasty Associated With Reason for Revision?
Status: Completed | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, rwpoolman, Professor Rudolf Wilhelm Poolman, Leiden University Medical Center
Other Study IDs: W.20.018)
Record Dates: First submitted 2021-05-03; First posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Osteo Arthritis Knee; Psychological Distress
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: • All patients undergoing primary total knee arthroplasty for osteoarthritis of the knee reported in the Dutch Arthroplasty Register.
  and
  • Patients who filled out the EQ-5D-3L anxiety/depression score.
  Interventions: Procedure: Knee Arthroplasty, knee revision arthoplasty

INTERVENTIONS:
Procedure: Knee Arthroplasty, knee revision arthoplasty — Primary knee arthroplasty (e.g., total, unicondylar and patellofemoral)

SUMMARY:
The aim of our study is to identify the influence of preoperative pain (NRS pain score and EQ5D pain score) and higher levels of anxiety and depression (EQ5D anxiety/depression score) and their interaction before primary total knee arthroplasty on revision surgery for unexplained symptoms after primary surgery.

DETAILED DESCRIPTION:
Knee arthroplasty can decrease pain and improve function in people with advanced osteoarthritis of the knee. It is a common procedure; over 25,000 primary knee arthroplasties are performed in the Netherlands each year[2]. A primary knee arthroplasty is defined as the first implantation of a prosthesis in the knee. Revision surgery is defined as any exchange (placement, replacement, or removal) or addition of 1 or more components of the prosthesis (e.g. patella resurfacing)[3]. About 12% of knee arthroplasties are revised within 10 years.

It is known that 1 in 5 patients rate themselves categorically dissatisfied after knee arthroplasty (the so-called unhappy knee). It seems sensible that the percentage of patients that has some dissatisfaction with their knee arthroplasty is likely much larger. After knee arthroplasty, some patients receive revision surgery based on clear reasons such as periprosthetic fracture and patellar dislocation, while in some patients that are dissatisfied revision surgery might be considered for less clear reasons such as a small technical issue, for a perceived technical issue, or with the idea that there is a low grade infection. Understanding the preoperative factors of postoperative pain and functional impairment, leading to dissatisfaction, may help to inform patients considering primary knee arthroplasty about the risk of revision surgery. Although pain and function of patients with higher preoperative pain scores before primary knee arthroplasty will improve as much as the scores of patients with lower preoperative pain scores, their final postoperative pain levels and function will remain inferior compared to patients with lower preoperative pain scores. Higher levels of anxiety and symptoms of depression before knee arthroplasty have also been related to worse postoperative patient reported outcome measures after surgery. Furthermore, the experience of pain and symptoms of depression are closely related to each other and they may influence each other in a bidirectional way. Determining the influence of preoperative pain and psychological distress (anxiety/depression) and their interaction on postoperative outcome seems to be crucial because mental and social health opportunities might be underdiagnosed and undertreated and the indication for a revision surgery may be based on a misdiagnosis of perceived or actual pathophysiology or technical deficiency in patients without a clear technical or medical indication for revision.

The aim of this study is to identify the influence of the preoperative pain (NRS pain score and EQ5D pain score) and higher levels of anxiety and depression (EQ5D anxiety/depression score) and their association before primary total knee arthroplasty (TKA) on revision surgery for unexplained symptoms after primary surgery.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing primary knee arthroplasty (e.g., total, unicondylar and patellofemoral) reported in the Dutch Arthroplasty Register.
* Patients who filled out the NRS pain score, EQ-5D 3L or EQ-5D 5L pain score or EQ-5D anxiety/depression score.

Exclusion Criteria:

* Other types of (revision) arthroplasty (hip / shoulder / ankle)
* Patients who did not fill out the NRS pain score, EQ-5D (3L or 5L) pain score or EQ-5D (3L or 5L) anxiety/depression score

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing primary knee arthroplasty (e.g., total, unicondylar and patellofemoral) reported in the Dutch Arthroplasty Register.
Sampling Method: Non-Probability Sample
Enrollment: 70754 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Revision surgery after knee arthroplasty | Duration until surgery, an average of 2.05 years.
  Our primary outcome measure was if a patient received revision surgery after knee arthroplasty (yes/no).
  We categorized the reason for revision in a consensus meeting among the investigators from this research group and experts in the Orthopaedic Surgery field into the following categories:
  * Clear reason for revision (patellar dislocation, insert wear, fracture, loosening and second stage revision after removal of knee arthroplasty)
  * Less clear reason for revision (infection, malalignment and instability)
  * Revision performed for unexplained symptoms without important pathophysiology (patellar pain, arthrofibrosis or progression of osteoarthritis (in case of unicondylar knee arthroplasty)).

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf Poolman, Prof, Principal Investigator — LUMC
Locations (1):
- LUMC, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No
We will derive data of patients undergoing primary knee arthroplasty from the Dutch Arthroplasty Register, the "Landelijke Registratie Orthopedische Implantaten" (LROI).
  We have submitted a research application to use data of the LROI for our study, which was judged by the "Wetenschappelijke Adviesraad" (WAR). After approval af the WAR, further agreements have been made between our research group and the LROI about the way in which the data were securely prepared. The specific dataset for our research question was prepared by the LROI and labeled by a specific research number (LROI2020-057 Poolman - Depressie en pijn bij KA). The LROI does not include names and addresses of patients. The citizen service number is encrypted by the LROI. The researchers will have no access to identifiable patient data.

REFERENCES:
- [Background] Carr AJ, Robertsson O, Graves S, Price AJ, Arden NK, Judge A, Beard DJ. Knee replacement. Lancet. 2012 Apr 7;379(9823):1331-40. doi: 10.1016/S0140-6736(11)60752-6. Epub 2012 Mar 6. PMID 22398175
- [Background] Spekenbrink-Spooren A, Van Steenbergen LN, Denissen GAW, Swierstra BA, Poolman RW, Nelissen RGHH. Higher mid-term revision rates of posterior stabilized compared with cruciate retaining total knee arthroplasties: 133,841 cemented arthroplasties for osteoarthritis in the Netherlands in 2007-2016. Acta Orthop. 2018 Dec;89(6):640-645. doi: 10.1080/17453674.2018.1518570. Epub 2018 Oct 23. PMID 30350747
- [Background] Labek G, Thaler M, Janda W, Agreiter M, Stockl B. Revision rates after total joint replacement: cumulative results from worldwide joint register datasets. J Bone Joint Surg Br. 2011 Mar;93(3):293-7. doi: 10.1302/0301-620X.93B3.25467. PMID 21357948
- [Background] Scott CE, Howie CR, MacDonald D, Biant LC. Predicting dissatisfaction following total knee replacement: a prospective study of 1217 patients. J Bone Joint Surg Br. 2010 Sep;92(9):1253-8. doi: 10.1302/0301-620X.92B9.24394. PMID 20798443
- [Background] Ferket BS, Feldman Z, Zhou J, Oei EH, Bierma-Zeinstra SM, Mazumdar M. Impact of total knee replacement practice: cost effectiveness analysis of data from the Osteoarthritis Initiative. BMJ. 2017 Mar 28;356:j1131. doi: 10.1136/bmj.j1131. PMID 28351833
- [Background] Tolk JJ, Waarsing JEH, Janssen RPA, van Steenbergen LN, Bierma-Zeinstra SMA, Reijman M. Development of Preoperative Prediction Models for Pain and Functional Outcome After Total Knee Arthroplasty Using The Dutch Arthroplasty Register Data. J Arthroplasty. 2020 Mar;35(3):690-698.e2. doi: 10.1016/j.arth.2019.10.010. Epub 2019 Oct 18. PMID 31711805
- [Background] Choi YJ, Ra HJ. Patient Satisfaction after Total Knee Arthroplasty. Knee Surg Relat Res. 2016 Mar;28(1):1-15. doi: 10.5792/ksrr.2016.28.1.1. Epub 2016 Feb 29. PMID 26955608
- [Background] van de Water RB, Leichtenberg CS, Nelissen RGHH, Kroon HM, Kaptijn HH, Onstenk R, Verdegaal SHM, Vliet Vlieland TPM, Gademan MGJ. Preoperative Radiographic Osteoarthritis Severity Modifies the Effect of Preoperative Pain on Pain/Function After Total Knee Arthroplasty: Results at 1 and 2 Years Postoperatively. J Bone Joint Surg Am. 2019 May 15;101(10):879-887. doi: 10.2106/JBJS.18.00642. PMID 31094979
- [Background] Bierke S, Haner M, Petersen W. Influence of somatization and depressive symptoms on the course of pain within the first year after uncomplicated total knee replacement: a prospective study. Int Orthop. 2016 Jul;40(7):1353-60. doi: 10.1007/s00264-015-3105-z. Epub 2016 Jan 28. PMID 26820743
- [Background] Bistolfi A, Bettoni E, Aprato A, Milani P, Berchialla P, Graziano E, Massazza G, Lee GC. The presence and influence of mild depressive symptoms on post-operative pain perception following primary total knee arthroplasty. Knee Surg Sports Traumatol Arthrosc. 2017 Sep;25(9):2792-2800. doi: 10.1007/s00167-015-3737-y. Epub 2015 Sep 21. PMID 26392343
- [Background] Duivenvoorden T, Vissers MM, Verhaar JA, Busschbach JJ, Gosens T, Bloem RM, Bierma-Zeinstra SM, Reijman M. Anxiety and depressive symptoms before and after total hip and knee arthroplasty: a prospective multicentre study. Osteoarthritis Cartilage. 2013 Dec;21(12):1834-40. doi: 10.1016/j.joca.2013.08.022. Epub 2013 Sep 4. PMID 24012622
- [Background] Ellis HB, Howard KJ, Khaleel MA, Bucholz R. Effect of psychopathology on patient-perceived outcomes of total knee arthroplasty within an indigent population. J Bone Joint Surg Am. 2012 Jun 20;94(12):e84. doi: 10.2106/JBJS.K.00888. PMID 22717836
- [Background] Konig HH, Born A, Gunther O, Matschinger H, Heinrich S, Riedel-Heller SG, Angermeyer MC, Roick C. Validity and responsiveness of the EQ-5D in assessing and valuing health status in patients with anxiety disorders. Health Qual Life Outcomes. 2010 May 5;8:47. doi: 10.1186/1477-7525-8-47. PMID 20444251
- [Background] Khatib Y, Jenkin D, Naylor JM, Harris IA. Psychological Traits in Patients Waiting for Total Knee Arthroplasty. A Cross-sectional Study. J Arthroplasty. 2016 Aug;31(8):1661-6. doi: 10.1016/j.arth.2016.01.053. Epub 2016 Feb 8. PMID 26944015
- [Background] Geisser ME, Roth RS, Theisen ME, Robinson ME, Riley JL 3rd. Negative affect, self-report of depressive symptoms, and clinical depression: relation to the experience of chronic pain. Clin J Pain. 2000 Jun;16(2):110-20. doi: 10.1097/00002508-200006000-00004. PMID 10870723
- [Background] Papakostidou I, Dailiana ZH, Papapolychroniou T, Liaropoulos L, Zintzaras E, Karachalios TS, Malizos KN. Factors affecting the quality of life after total knee arthroplasties: a prospective study. BMC Musculoskelet Disord. 2012 Jun 29;13:116. doi: 10.1186/1471-2474-13-116. PMID 22748117
- [Background] Riddle DL, Jiranek WA, Hayes CW. Use of a validated algorithm to judge the appropriateness of total knee arthroplasty in the United States: a multicenter longitudinal cohort study. Arthritis Rheumatol. 2014 Aug;66(8):2134-43. doi: 10.1002/art.38685. PMID 24974958